CLINICAL TRIAL: NCT03695874
Title: Development of a Quality of Life Measurement Scale in Hereditary Haemorrhagic Telangiectasia (HHT) Disease.
Acronym: ELECT-RO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0543
Record Dates: First submitted 2018-09-30; First posted 2018-10-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: statistical purification: 400 Hereditary Haemorrhagic Telangiectasia patients:
  * over 18 years
  * able to read French
  * with clinically confirmed Hereditary Haemorrhagic Telangiectasia disease (presence of at least 3 Curaçao criteria) and / or molecular biology
  * who received the information and did not object to participate in the study
  Interventions: Other: Phase 1 : fill out 1 scale
- Phase 2: statistical validation: 200 Hereditary Haemorrhagic Telangiectasia patients:
  * over 18 years
  * able to read French
  * with clinically confirmed Hereditary Haemorrhagic Telangiectasia disease (presence of at least 3 Curaçao criteria) and / or molecular biology
  * who received the information and did not object to participate in the study
  Interventions: Other: Phase 2 : fill out 1 scale and 4 questionnaires

INTERVENTIONS:
Other: Phase 1 : fill out 1 scale — Patients will be asked to complete questionnaires.
  Group 1: the purpose is to simplify a 75 items scale by a statistical analysis of the data collected from 400 patients. The statistical purification will allow to finalize an abbreviated scale (20-25 items).
  Doctors specialized in Hereditary Haemorrhagic Telangiectasia may suggest that patients enter the study. After submission of the information notice and collection of their non-opposition, patients will have the choice to fill out the paper version or the electronic version of the scale and questionnaires.
  Groups: Phase 1: statistical purification
Other: Phase 2 : fill out 1 scale and 4 questionnaires — Patients will be asked to complete questionnaires.
  Group 2: the purpose is to validate the abbreviated scale by a statistical analysis of the data collected from 200 patients. The statistical validation will allow to check the consistency and correlation of the abbreviated scale with other scales: a general Quality Of Life scale (SF36), an anxiety and depression scale (HAD), a social support scale (SSQ6) and a scale of regulation emotional (CERQ) and to test and re-test to check fidelity of the abbreviated scale.
  Doctors specialized in Hereditary Haemorrhagic Telangiectasia may suggest that patients enter the study. After submission of the information notice and collection of their non-opposition, patients will have the choice to fill out the paper version or the electronic version of the scale and questionnaires.
  Groups: Phase 2: statistical validation

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT) is a rare inherited genetic disease of autosomal dominant inheritance with a prevalence of 1/6000. It is manifested by haemorrhages, mucocutaneous telangiectasias and visceral arteriovenous malformations. These symptoms significantly affect the daily lives of patients, their social relationships and their working lives.

HAS (Haute Autorité de Santé) national recommendations focus on assessing and improving the quality of life (QOL) of patients. Many scales for measuring QOL exist but they are most often general and therefore have the disadvantage of not taking into account the particularities of pathologies and their symptoms and do not allow to have a precise vision of their impact on QOL.

It is important to be able to evaluate this impact, to determine its nature and to quantify it so that health professional can adapt their proposal for the management of HHT patients. And only the development of a specific and validated QOL measurement scale will allow them to access this information.

The aim of this study is to develop a scale of measurement of quality of life in HHT disease and to validate it, a scale specific to HHT, simple and fast to fill by the patients themselves.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* able to read French
* with clinically confirmed Hereditary Haemorrhagic Telangiectasia disease (presence of at least 3 Curaçao criteria) and / or molecular biology
* who received the information and did not object to participate in the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an Hereditary Haemorrhagic Telangiectasia disease.
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Validity of the factor structure of the developed measurement scale. | 1 hour
  Saturation coefficients of the exploratory factor analysis observed on the sample of 400 participants, confirmatory factor analysis (CFA) adjustment indices on the sample of 200 participants, and factorial weights observed on the AFC will be combined to evaluate the structural validity of the measurement scale.
Validity of the reliability of the developed measurement scale. | 1 hour
  Cronbach alphas coefficients, composite reliability values (rho) and percentages of extracted variance will be combined to assess the Reliability of the measurement scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence pour la Maladie de Rendu-Osler - Service de Génétique Clinique - HOSPICES CIVILS DE LYON - Groupement Hospitalier Est, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le TTT, Martinent G, Dupuis-Girod S, Parrot A, Contis A, Riviere S, Chinet T, Grobost V, Espitia O, Dussardier-Gilbert B, Alric L, Armengol G, Maillard H, Leguy-Seguin V, Leroy S, Rondeau-Lutz M, Lavigne C, Mohamed S, Chaussavoine L, Magro P, Seguier J, Kerjouan M, Fourdrinoy S. Development and validation of a quality of life measurement scale specific to hereditary hemorrhagic telangiectasia: the QoL-HHT. Orphanet J Rare Dis. 2022 Jul 19;17(1):281. doi: 10.1186/s13023-022-02426-2. PMID 35854330